CLINICAL TRIAL: NCT02712723
Title: Femara (Letrozole) Plus Ribociclib (LEE011) or Placebo as Neo-adjuvant Endocrine Therapy for Women With ER-positive, HER2-negative Early Breast Cancer
Brief Title: Letrozole Plus Ribociclib or Placebo as Neo-adjuvant Therapy in ER-positive, HER2-negative Early Breast Cancer
Acronym: FELINE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qamar Khan (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Qamar Khan, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLEE011XUS10T
Record Dates: First submitted 2016-02-25; First posted 2016-03-18 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer
Keywords: ER+, HER2-negative breast cancer; Stage II or III; Letrozole; Femara; Ribociclib; LEE011; Neo-adjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; ribociclib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo + Letrozole (Active Comparator): Placebo randomized to 3 capsules/day 3 weeks on/1week off or 2 capsules/day continuous dosing + Letrozole 2.5 mg PO daily
  Interventions: Drug: Letrozole; Drug: Placebo
- Ribociclib 600 mg + Letrozole (Experimental): Ribociclib 600 mg PO daily 21 days on/7 days off + Letrozole 2.5 mg PO daily
  Interventions: Drug: Letrozole; Drug: Ribociclib
- Ribociclib 400 mg + Letrozole (Experimental): Ribociclib 400 mg continuous daily dosing + Letrozole 2.5 mg PO daily
  Interventions: Drug: Letrozole; Drug: Ribociclib

INTERVENTIONS:
Drug: Letrozole — Nonsteroidal aromatase inhibitor
  Other Names: Femara; CGS 20267; LTZ
Drug: Ribociclib — Oral cyclin-dependent kinase (CDK) inhibitor
  Other Names: LEE011; LEE-011
  Arms: Ribociclib 400 mg + Letrozole; Ribociclib 600 mg + Letrozole
Drug: Placebo — Placebo for ribociclib
  Arms: Placebo + Letrozole

SUMMARY:
The purpose of this study is to determine if ribociclib in combination with letrozole for 24 weeks as neoadjuvant endocrine therapy increases the proportion of women with Pre-operative Endocrine Prognostic Index (PEPI) score of 0 at surgery compared to patients treated with letrozole alone therefore allowing more patients excellent outcomes without chemotherapy.

DETAILED DESCRIPTION:
Subjects will be randomized (1:1:1) to either letrozole plus placebo vs. letrozole plus continuous dosing of ribociclib vs. letrozole plus intermittent dosing (3-weeks-on/1-week-off) of ribociclib.

The difference in clinical, pathologic and radiologic response as well as Pre-operative Endocrine Prognostic Index (PEPI) scores across the three treatments arms will be examined. Subjects will also be followed for 5 years post-treatment to determine if ribociclib in combination with letrozole for 24 weeks results in improved 5 year Relapse Free Survival (RFS) compared to letrozole alone.

ELIGIBILITY:
Key Inclusion Criteria:

* Pathologically confirmed invasive breast cancer by core needle biopsy
* Female subjects, age ≥ 18 years
* Only postmenopausal women will be eligible.
* Performance Status: Eastern Cooperative Oncology Group (ECOG) score 0-2
* Invasive breast cancer must be ER+ in ≥66 % of the cells or ER Allred score 6-8
* Invasive breast cancer must be HER2 negative.
* Clinical Stage II or III (by clinical measurement and/or breast imaging)

Key Exclusion Criteria:

* Subjects meeting any of the exclusion criteria at baseline will be excluded from study participation.
* Current use of other investigational agents
* Inflammatory breast cancer defined as clinically significant erythema of the breast and/or documented dermal lymphatic invasion (not direct skin invasion by tumor or peau d'orange without erythema)
* An excisional biopsy of this breast cancer
* Surgical axillary staging procedure prior to study entry
* Hormone replacement therapy of any type, megestrol acetate, or raloxifene within four weeks prior to first study treatment
* Clinical or radiographic evidence of metastatic disease
* Clinically significant, uncontrolled heart disease
* Herbal preparations/medications as listed in Appendix B of the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Rate of Pre-operative Endocrine Prognostic Index (PEPI) score 0 at surgery between ribociclib containing arms (combined) vs letrozole alone arm | At Surgery (22 weeks)

SECONDARY OUTCOMES:
Rate of complete cell cycle arrest at 2 weeks between ribociclib containing arms (combined) vs letrozole alone arm: Complete cell cycle arrest is defined as Ki67 at day 14 of < 2.7% | Day 14 of Cycle 1
Pathologic complete response rate (pCR rate): pCR rate is defined as the proportion of patients with no histologic evidence of invasive tumor cells in the surgical breast specimen and the axillary lymph nodes | At Surgery (Days 8-15 of Cycle 6)
Clinical complete response rate (cCR rate): cCR rate is defined as the proportion of patients with no residual tumor by clinical exam | Post-surgery (Once in the first 4 weeks of post-op, then once every 6 months for 5 years post-op)
5 Year Relapse Free Survival (RFS) | 5 years post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Qamar Khan, MD, Principal Investigator — University of Kansas Medical Center
Locations (13):
- United States (13):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - Cancer Research Collaboration, Santa Ana, California
  - University of Miami Sylvester Comprehensive Cancer Center, Deerfield Beach, Florida
  - University of Kansas Cancer Center - West, Kansas City, Kansas
  - University of Kansas Cancer Center - Overland Park, Overland Park, Kansas
  - University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Kansas Cancer Center - South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Columbia University Medical Center, New York, New York
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No